CLINICAL TRIAL: NCT05212116
Title: A Phase Ib, Exploratory, Double Blind, Placebo Controlled, Parallel Group, Study of SDI-118 to Evaluate Safety, Tolerability, and Pharmacodynamics Including Cognitive Function in Male and Female Participants in Remission From Depression
Brief Title: A Study of SDI-118 in Participants in Remission From Depression
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Development Plan Amended
Sponsor: Syndesi Therapeutics (Industry)
Collaborators: P1vital Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYND004; 2020-003748-10 (EudraCT Number)
Record Dates: First submitted 2021-05-26; First posted 2022-01-27 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Depression in Remission
Keywords: Depression; Major Depressive Disorder; Depression in Remission
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Intervention Model: Parallel Assignment Masking: Double Blind Primary Purpose: Treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SDI-118 low dose (Experimental): SDI-118 (low dose) orally once daily (QD) for 17±1 day.
  Interventions: Drug: SDI-118
- SDI-118 high dose (Experimental): SDI-118 (high dose) orally once daily (QD) for 17±1 day.
  Interventions: Drug: SDI-118
- Placebo (Placebo Comparator): Placebo orally once daily (QD) for 17±1 day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SDI-118 — SDI-118 is presented as low dose, and high dose capsules.
  Arms: SDI-118 high dose; SDI-118 low dose
Drug: Placebo — The Matching Placebo for SDI-118 is mannitol in capsules.
  Arms: Placebo

SUMMARY:
This is a multi-center, double-blind, randomized, placebo-controlled study to determine the safety, tolerability, and pharmacodynamics of SDI-118 in a once daily (QD) dosing regimen on male and female study participants reporting with cogntive decline and who in remission from depression.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between 25 and 55 years of age (inclusive) at screening.
* Are remitted from depression.
* Have received prescribed treatment with an antidepressant or a recognised psychotherapy for depression (e.g. cognitive behaviour therapy) for a previous MDE
* Report present subjective cognitive impairment (such as difficulty concentrating, slow thinking, and difficulty in learning new things or remembering things).
* Have not been treated with antidepressants or received other psychotherapy for depression for at least six weeks prior to Screening Visit 1.
* Otherwise healthy with no clinically significant abnormalities as determined by medical history, physical examination, blood chemistry assessments, haematologic assessments, and urinalysis, measurement of vital signs, and Electrocardiogram (ECG).
* Negative serology test for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies at screening.
* Have a body mass index (BMI) of 18 to 36 inclusive.
* Agree not to use herbal medications (including herbal tea, St. John's Wort), within 14 days prior to study agent administration through to the final follow-up visit.
* Participants must be able and willing to give written, informed consent, indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* The participant, in the opinion of the investigator, is willing and able to adhere to the study visit schedule and other requirements, prohibitions and restrictions of the study.

Exclusion Criteria:

* They are left-handed.
* Have immediate recall of greater than 22 words from the International Shopping List Test (ISLT) and have delayed recall of greater than 8 words from the ISLT 15 mins after the presentation of the word list.
* Positive urine drug screen or alcohol breath test at screening or assessment visits.
* History or presence of significant neurological or psychiatric conditions except those related to MDD.
* Any suicidal ideation of type 4 or 5 in the Columbia Suicide Severity Rating Scale (C-SSRS) in the past 3 months prior to screening or at screening or baseline visit.
* Has a known clinically relevant structural brain abnormality as determined by e.g. previous MRI, or, persistent MRI imaging artefact which is judged to produce extensive imaging distortions.
* Has a disease or takes medication that could, in the investigator's and/or sponsor's opinion, interfere with the assessments of safety, tolerability, or efficacy, or interfere with the conduct or interpretation of the study.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | 17 days
  Adverse events (AEs) will be coded using medical dictionary for regulatory activities (MedDRA). An AE is any untoward medical occurrence in a participant administered a study drug and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medical product whether or not considered related to the medical product. An AE is considered "serious" if, in the view of either the investigator or sponsor, the event: results in death, is life-threatening, results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, results in congenital anomaly or birth defect, requires hospitalization or prolongation to hospitalization, or other medically important event.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | 17 days
  Number of participants with potentially clinically significant laboratory values (hematology/chemistry/urinalysis)
Number of participants with vital sign abnormalities and/or adverse events (AEs) | 17 days
  Number of participants with potentially clinically significant vital sign values
Number of participants with routine 12 lead electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) | 17 days
  Number of participants with potentially clinically significant ECG values
Number of participants with C-SSRS abnormalities and/or Adverse Events (AEs) | 17 days
  Number of participants with potentially clinically significant changes in C-SSRS values.
Number of participants with routine physical examination abnormalities and/or Adverse Events (AEs) | 17 days
  Number of participants with potentially clinically significant changes in physical examination.
Number of participants with Changes in the Cogstate Brief Battery, including abnormalities and/or Adverse Events (AEs) | 17 days
  Number of participants with potentially clinically significant changes in the Cogstate Brief Battery values
Number of participants with Changes in the Digital Symbol Substitution Test, including abnormalities and/or Adverse Events (AEs) | 17 days
  Number of participants with potentially clinically significant changes in the DSST values.
Number of participants with Changes in the Controlled Oral Word Association Test, including abnormalities and/or Adverse Events (AEs) | 17 days
  Number of participants with potentially clinically significant changes in the COWAT values.
Number of participants with Changes in the Category Fluency Test, including abnormalities and/or Adverse Events (AEs) | 17 days
  Number of participants with potentially clinically significant changes in the CFT values.

SECONDARY OUTCOMES:
Changes in Blood Oxygen Level Dependent (BOLD) signal | 17 days
  As measured by changes in deoxyhemoglobin levels driven by localized changes in brain blood flow and blood oxygenation in brain networks associated with executive function (working memory), including the prefrontal cortex, the hippocampus, and the associated limbic networks, during performance of the N-Back Tasks
Changes in Blood Oxygen Level Dependent (BOLD) signal | 17 days
  As measured by changes in processing of emotional stimuli during theperformance of the FEP task.
Performance measures associated with executive function (working memory) during the N-Back Tasks | 17 days
  As measured by both response accuracy and response latency between cue stimulus and detection of this cue in the presented trial stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Smith, DM, Principal Investigator — University of Oxford; Maeve Duffy, PhD, Study Chair — Syndesi Therapeutics
Locations (3):
- United Kingdom (3):
  - University of Manchester, Manchester, Lancashire
  - University of Oxford, Oxford, Oxfordshire
  - Cardiff University, Cardiff, Wales

IPD SHARING:
Plan to Share IPD: No